CLINICAL TRIAL: NCT02971878
Title: Adding Antioxidants Into Human Embryo Culture Media
Brief Title: Comparisons of Human Embryonic Development Using Single Medium With and Without the Addition of Antioxidants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertilitetscentrum AB (Other)
Collaborators: Vitrolife (Industry)
Responsible Party: Principal Investigator, Thorir Hardarson, Laboratory Director, Fertilitetscentrum AB
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GTL-X
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Culture Media; Blastocyst; Antioxidants; Embryo; Human
MeSH Terms: interventions — Acetylcarnitine; allantoicase; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Culture media without addition of antioxidants
- Treatment (Active Comparator): Culture media with the addition of antioxidants
  Interventions: Biological: Acetyl-L-carnitine (ALC), N-acetyl-L-cysteine (NAC) and α-lipoic acid (ALA)

INTERVENTIONS:
Biological: Acetyl-L-carnitine (ALC), N-acetyl-L-cysteine (NAC) and α-lipoic acid (ALA) — Human embryos will be cultured in media that contains 3 antioxidants (Acetyl-L-carnitine (ALC), N-acetyl-L-cysteine (NAC) and α-lipoic acid (ALA)) that can be found in the in vivo Environment.
  Arms: Treatment

SUMMARY:
Aim: To investigate the impact of antioxidants (acetyl-L-carnitine, N-acetyl-L-cysteine and a-lipoic acid) on embryo development and subsequently the clinical outcome. Including clinics using low oxygen and ambient air during embryo culture. Analysed with time-lapse system.

Study media: G-TL with antioxidants. Control media: Same media without antioxidants. Type of study: Study comparing blastocyst development on the same cohort of oocytes using two different media, G-TL versus G-TL supplemented with antioxidants. Statistics based on an absolute increase in Good Quality Blastocysts on day 5 of 7%.

Design: Multicentre prospective randomized sibling trial. Single blastocyst transfer. Superiority study Primary Endpoint: Good Quality Blastocysts on day 5 per allocated normally fertilized oocyte.

Patients: Comparative embryo sibling study with 128 patients included.

DETAILED DESCRIPTION:
Study objective: Study comparing blastocyst development on the same cohort of oocytes using two different media, G-TL versus G-TL supplemented with antioxidants.

Primary endpoint: Percentage of good quality blastocysts (GQB) per fertilized oocyte on day 5.

Secondary endpoints

* Embryo development day 3, 5 and 6
* Embryo quality day 3, 5 and 6
* Total blastocyst formation (day 5 and day 6)
* Utilization rate (embryos available for transfer and cryopreservation)
* Implantation rate
* Clinical pregnancy rate

Setup: Prospective embryo sibling, superiority study

MATERIALS AND METHODS Intervention New type of embryo culture media used for in vitro culture of human IVF embryos.

Power analysis The planning and the power analysis was made together with a statistician, Nils-Gunnar Pehrsson.

From retrospective data using simulation, the intra individual SD for the difference in % GQB between the two media strategies was estimated to 32%. In order to find a difference in 8% in GQB between the two media with power 80% with paired T-test 128 couples will be needed.

Randomization Couples will be enrolled in the study after fertilization check (day 1). A minimum of 6 zygotes is required for participation.

Stratified randomization of the zygotes by couple will be performed. For each couple the zygotes will be numbered.

These zygotes for each couple will then be block (by two) randomized to the two media types; A (Traditional culture media = Control) and B (Antioxidant media = intervention). In both groups traditional culture will be performed. Allocation will be performed in a 1:1 ratio according to a unique randomization list for each couple.

Blinding To minimize possible bias for the primary outcome (GQE D5) the embryologist performing the morphological evaluation on day 5/6 will not know which group the embryos belong to.

Both the physician and the couple will be blinded to which group they have been allocated.

IVF treatment procedure A traditional IVF treatment will be performed including ovarian stimulation and oocyte pick-up using the standard methods at the clinics.

Embryo assessment and timing of assessment according to Alpha/ESHRE consensus criteria.

Morphological scoring Blastocyst morphology will be scored according to Consensus Scoring system for blastocysts (Istanbul Consensus workshop on embryo assessment) and the morphology will be documented with individual photos of each blastocyst. Blastocyst scoring will be performed under an inverted microscope on day 5 and day 6. A good quality blastocyst is defined as at least Grade 2:2:2 according to Istanbul Consensus grading system. (Balaban et al., 2011).

DOCUMENTATION All patients participating in the study will be documented on a computerized CRF. This document will be related to patients' records with all relevant clinical and laboratory data from the specific IVF cycle. Through the journal system (WinIVF) used at Fertilitetscentrum, it will be possible to generate a complete list of all the variables included in the study.

Patients who have been asked to participate in the study but did not fulfill the criteria for randomization will also be registered.

STATISTICAL ANALYSIS Both an Intention-to-Treat (ITT) population and a Per Protocol (PP) population will be defined. Primary efficacy variable in this superiority study will be difference in %GQB between the two media types for each couple. Primary statistical analysis will be two-sided paired T-test regarding the mean of difference in %GQB between Standard culture media and Antioxidant media on the ITT population. A two sided 95% confidence interval for the mean difference in %GOB between the two media will be calculated. All significance tests will be two-sided and conducted at the 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Couples with female, male or unexplained infertility intending to undergo IVF
* The couple should have received verbal and written information/consent about the study.
* 6 or more fertilized oocytes on day 1
* Blastocyst culture and transfer on day 5
* Signed written consent

Exclusion Criteria:

* Previous participation in the study.
* Testicular biopsy patients (TESA/TESE)
* Fewer than 6 fertilized oocytes.
* If split IVF is needed.
* Total freeze on day 3

Ages: 20 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of good quality blastocysts (GQB) per randomized embryo | 7 months

SECONDARY OUTCOMES:
Pregnancy rate | 10 months
Utilization rate | 7 months
Embryo development (Kinetics) day 3,5 & 6 | 7 months
Implantation rate | 8 months
Embryo quality dag 3,5 and 6 | 7 months
Total blastocyst rate | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Thorir Hardarson, PhD, Study Chair — Fertilitetscentrum AB
Locations (1):
- Fertilitetscentrum, Gothenburg, Box 5418, Sweden